CLINICAL TRIAL: NCT03082872
Title: Randomized Comparison Between Cemented K-wire Fixation vs Open Transfixion Pinning for the Treatment of Shaft Fractures of Middle Phalanges
Brief Title: Cemented K-wire Fixation vs Open Transfixion Pinning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THHMU201763
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Closed Fracture of Finger; Finger Fracture
Keywords: Reduction, Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Patients with middle proximal fractures of fingers
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cemented K-wire Fixation (Experimental): Fractures were transverse (n=32), short oblique or spiral (n=5), and comminuted (n=14) fractures.
  Interventions: Device: Cemented K-wire; Device: Transfixion Pinning
- Open Transfixion Pinning (Experimental): Fractures were transverse (n=28), short oblique or spiral (n=4), and comminuted (n=15) fractures.
  Interventions: Device: Cemented K-wire; Device: Transfixion Pinning

INTERVENTIONS:
Device: Cemented K-wire — Fracture of proximal phalanx was treated with Cemented K-wire.
Device: Transfixion Pinning — Fracture of proximal phalanx was treated with transfixion pinning.

SUMMARY:
To introduce a novel external-fixation technique using the combination of K-wires and cement, and the objective of this report is also to compare the technique with conventional open transfixion pinning.

DETAILED DESCRIPTION:
Shaft fractures of the middle phalanx are common injuries that are often difficult to treat. Currently, fracture fixation is usually achieved by using K-wire, but pin configurations are controversial.The objective of this report is to introduce treatment of shaft fractures of middle phalanx with a novel external-fixation technique using combined K-wires and cement. For comparison, we also included another group of patients who were treated using open transfixion pinning.A total of 98 patients (98 fingers) with shaft fractures of middle phalanx were randomly allocated to group A (n=51) and B (n=47). Fingers in group A were treated with cemented K-wire fixation, and fingers in group B were treated using conventional open transfixion pinning. Time of bone healing, range of motion of the fingers, and joint motion were assessed. A p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patient aged between 18 and 65 years;
* acute fractures within 15 days;
* closed fractures or fractures with small open wound less than 1.5 cm;
* involvement of single middle phalanges of index to little fingers;
* shaft fractures; at least 5 mm in length of the most distal and proximal fragments so that K-wires can be secured;
* transversal, short oblique or spiral fractures;
* comminuted fractures of middle third phalanx;
* normal opposite hand for comparison.

Exclusion Criteria:

* patients younger than 18 years are excluded because of skeletal immaturity;
* patients older than 65 years are excluded because of possible osteoporosis;
* multiple finger involvement; severe open injury or crush injuries;
* combined tendon or neurovascular injuries; involvement of articular surface;
* old fractures exceeding 15 days because close reduction most likely became difficult;
* combined tendon, nerve, or artery injuries or diseases;
* diabetes, gout, ganglion;
* osseous tumors, and other disease affecting bony structures and joint motion;
* patients who declined to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Bone healing | Up to 12 weeks. From date of randomization until the date of first documented progression from any cause, which is assessed up to 12 weeks.
  Time of bone healing

SECONDARY OUTCOMES:
Joint motion | Up to 2 years. From date of randomization until the date of second documented progression from any cause, which is assessed up to 2 years.
  Range of motion of MCP, PIP, and DIP joints

OTHER OUTCOMES:
Patient satisfaction | Up to 2 years. From date of randomization until the date of third documented progrssion from any cause, which is assessed up to 2 years.
  Patient self assessment based on 100-mm visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No
No plan to share the IPD data

REFERENCES:
- [Result] Edwards GS Jr, O'Brien ET, Heckman MM. Retrograde cross-pinning of transverse metacarpal and phalangeal fractures. Hand. 1982 Jun;14(2):141-8. doi: 10.1016/s0072-968x(82)80005-3. No abstract available. PMID 7117927
- [Result] Margic K. External fixation of closed metacarpal and phalangeal fractures of digits. A prospective study of one hundred consecutive patients. J Hand Surg Br. 2006 Feb;31(1):30-40. doi: 10.1016/j.jhsb.2005.09.013. Epub 2005 Nov 15. PMID 16293357
- [Result] Gaston RG, Chadderdon C. Phalangeal fractures: displaced/nondisplaced. Hand Clin. 2012 Aug;28(3):395-401, x. doi: 10.1016/j.hcl.2012.05.032. Epub 2012 Jun 26. PMID 22883890